CLINICAL TRIAL: NCT01953523
Title: Clinical Intervention Study: Adverse Events and Clinical Outcomes for the Deployment of Adipose Derived SVF (Rich in Adult Stem Cells and Growth Factors)for Select Orthopedic, Neurologic, Urologic, and Cardio-Pulmonary Conditions.
Brief Title: Safety and Clinical Outcomes Study: SVF Deployment for Orthopedic, Neurologic, Urologic, and Cardio-pulmonary Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elliot Lander (Industry)
Responsible Party: Sponsor-Investigator, Elliot Lander, Medical Director, Cell Surgical Network Inc.
Organization: Cell Surgical Network Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSN111
Record Dates: First submitted 2013-09-02; First posted 2013-10-01 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Neurodegenerative Diseases; Osteoarthritis; Erectile Dysfunction; Autoimmune Diseases; Cardiomyopathies; Emphysema
Keywords: erectile dysfunction; peyronies; interstitial cystitis; cardiomyopathy; emphysema; copd; arthritis; multiple sclerosis; parkinson's
MeSH Terms: conditions — Neurodegenerative Diseases; Osteoarthritis; Erectile Dysfunction; Autoimmune Diseases; Cardiomyopathies; Emphysema; Cystitis, Interstitial; Pulmonary Disease, Chronic Obstructive; Arthritis; Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deployment of stromal vascular fraction (Experimental): Administration of autologous adipose derived SVF
  Interventions: Procedure: Administration of autologous adipose derived SVF

INTERVENTIONS:
Procedure: Administration of autologous adipose derived SVF — Intra-venous, intra-articular, and soft tissue injection delivery of SVF

SUMMARY:
To evaluate for any adverse effects that may be related to the administration and reception of autologous adipose derived stromal vascular fraction (SVF). Secondarily, the study monitors the results of subjective and objective findings as it applies to the non-blinded deployment of autologous SVF for various inflammatory and/or degenerative conditions including select orthopedic, neurologic, urologic and cardio-pulmonary conditions. SVF deployments include intra-venous, intra-articular, and soft tissue injections.

DETAILED DESCRIPTION:
SVF Stromal Vascular Fraction is obtained by lipoharvesting, procurement, and lipo-transfer as a same day operative procedure

ELIGIBILITY:
Inclusion Criteria

* Patient must be age 16 or older
* Patient must have a degenerative disease or inflammatory disease that meets criteria for treatment under the IRB which includes: Arthritis, Auto-immune disease,COPD, Cardiomyopathy, Peyronies Disease,Interstitial Cystitis, Erectile Dysfunction, and Neurodegenerative disease such as Parkinsons, ALS, Neuropathy.
* Patient must be healthy enough to tolerate a local anesthetic

Exclusion Criteria:

* Patient must not have active cancer
* Patient must not have active infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Outcome measures will include the number of participants with adverse events related to either SVF deployment or the lipo-harvesting procedure.

SECONDARY OUTCOMES:
Changes in the Oswestry Disability Index | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the Oswestry Disability Index Score will be measured. Outcomes represent changes from baseline in symptom and abilities scores on 11 questions.
Changes in the Neck Disability Index | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the Neck Disability Index Score will be measured. Outcomes represent changes from baseline in symptom and abilities scores on 10 questions.
Changes in Koos Physical Function Shortform | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in Koos Physical Function Shortform will be measured. Outcomes represent changes in level of function score from none to extreme.
Changes in Hoos Physical Function Shortform | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in Hoos Physical Function Shortform will be measured. Outcomes represent changes in level of function score from none to extreme.
Changes in the DASH questionnaire | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the DASH Questionnaire Score will be measured. Outcomes represent changes from baseline in symptoms and abilities scores on 11 questions.
Changes in the Visual Analog Pain Score | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the Visual Analog Pain Score will be measured. Outcomes represent changes from baseline from none to severe.
Changes in the Aqol-4 | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the Aqol-4 Assessment of Quality of Life Instrument will be measured. Outcomes represent changes from baseline in 12 subjective scores.
Changes in the O'leary-Sant IC Questionnaire | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the O'leary-Sant IC Questionnaire will be measured. Outcomes represent changes from baseline in 8 symptom and problem scores
Changes in PUF Symptom Scale | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the PUF Symptom Scale will be measured. Outcomes represent changes from baseline in in 8 symptom and bother scores.
Changes in the IIEF Questionnaire | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the IIEF Questionnaire Score will be measured. Outcomes represent changes in erectile function from baseline in 5 sexual function scores.
EHGS Grading Score measuring change in hardness score | Outcome measures will be evaluated at baseline, 3,6,9,12,15,18,21,24,27,30,33,36 months. Outcomes tests will be given yearly after 36 months for an average time frame of 5 years and estimated time frame maximum of 10 years.
  Changes in the EHGS Grading Score will be measured. Outcomes represent changes from baseline in erection hardness on a scale of 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Berman, MD, Principal Investigator — Cell surgical network
Locations (1):
- California Stem Cell Treatment Center, Rancho Mirage, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Finishing 1000 patient safety paper for peer review and publication.

REFERENCES:
- [Derived] Khera M, Albersen M, Mulhall JP. Mesenchymal stem cell therapy for the treatment of erectile dysfunction. J Sex Med. 2015 May;12(5):1105-6. doi: 10.1111/jsm.12871. No abstract available. PMID 25974235
- See also: cell surgical network — http://www.stemcellrevolution.com